CLINICAL TRIAL: NCT05718089
Title: Individual Responses in Insulin Sensitivity to Different Exercise Modalities in Persons With Overweight: a Randomized Cross-over Pilot Study
Brief Title: Precision Exercise Therapeutics (PET-pilot)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Cody Garett Durrer, PhD. Postdoc, Rigshospitalet, Denmark
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: H-22040452
Record Dates: First submitted 2023-01-17; First posted 2023-02-08 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Overweight; Healthy
MeSH Terms: conditions — Overweight | interventions — High-Intensity Interval Training; Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Participants will be randomly allocated, following successful completion of the baseline measurements. An independent statistician generates a computer-generated randomization schedule including six possible sequence orders using balanced blocks, stratified by sex.
  The schedule will be forwarded to a secretary not involved in any study procedures and will be stored on a password-protected computer. Sequentially numbered (according to the sequence) opaque, sealed envelopes will be prepared and stored in a locked cabinet in an access restricted room. The envelopes will be lined with aluminum foil to render the envelope impermeable to light. Following the baseline measurements, a study nurse, not involved with any study procedures, will open the envelope, and inform the researcher about the order. The participant be informed about the trial condition upon arrival to lab for the experiments (i.e. on the first morning of each set of trial conditions).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Continuous aerobic exercise (Experimental): The participants will complete a 10-min warm up, followed by 40 min of continuous aerobic exercise at an individualized intensity at 64-76% of the maximal heart rate HRmax on a bicycle ergometer/walking.
  Interventions: Other: Continuous aerobic exercise
- High intensity interval training (Experimental): The training consists of 10 minutes of warm up followed by 25 minutes of high intensity interval training (5 bouts of 4 min at >85% HRmax interspaced by 4 minutes of low intensity training) and finally a 4 min cool-down.
  Interventions: Other: High intensity interval training
- Resistance training (Experimental): The participants will complete moderate intensity whole-body resistance training. This will consist of 4 sets with 4 exercises (leg press, chest press, back row, leg extension in appropriate machines) with a brief warm-up prior to each exercise. Each set will be interspersed by 2-min breaks. Each set (including breaks) will thus equate to 2.5 min. Intensity will be set a 12-repetition max (RM, i.e., can repeated no more than 12 times) or 10 repetitions with 1-2 repetitions in reserve (i.e., 10 repetitions where failure would occur within 1-2 more repetitions).
  Interventions: Other: Resistance training

INTERVENTIONS:
Other: Continuous aerobic exercise — The "Continuous aerobic exercise" session will be performed in total two times, as it will be repeated in sets on consecutive weeks (e.g. Two Tuesdays in a row) with a 1-week wash-out period. The " Continuous aerobic exercise" intervention is matched to the other arms on the time spend for each bout equating a total of 50 minutes of exercise per session.
  An oral glucose tolerance test will be performed 24 hours and 48 hours after the exercise bout.
  Arms: Continuous aerobic exercise
Other: High intensity interval training — The "High intensity interval training" session will be performed in total two times, as it will be repeated in sets on consecutive weeks (e.g. Two Tuesdays in a row) with a 1-week wash-out period. The "High intensity interval training" intervention is matched to the other arms on the time spend for each bout equating a total of 50 minutes of exercise per session.
  An oral glucose tolerance test will be performed 24 hours and 48 hours after the exercise bout.
  Arms: High intensity interval training
Other: Resistance training — The "Resistance training" session will be performed in total two times, as it will be repeated in sets on consecutive weeks (e.g. Two Tuesdays in a row) with a 1-week wash-out period. The "Resistance training" intervention is matched to the other arms on the time spend for each bout equating a total of 50 minutes of exercise per session.
  An oral glucose tolerance test will be performed 24 hours and 48 hours after the exercise bout.
  Arms: Resistance training

SUMMARY:
The aim of this randomized cross-over study is to collect information for the design of a precision exercise therapy cohort that will predict what modality of physical activity a physically inactive individual with overweight should perform to increase insulin sensitivity given their unique biology, environment, and context.

DETAILED DESCRIPTION:
This pilot study is needed prior to launching precision therapeutics programs, with the purpose to decrease the risk of research waste, increase the reliability of the experimental tests and estimate adequate sample size.

25 participants will be recruited to undergo three sets of experiments. An experiment consists of one exercise bout followed by an assessment of whole-body insulin sensitivity (measured from a oral glucose tolerance test) 1 and 2 days following the completion of the exercise bout yielding 19 study days of 3 hours each across 7 weeks, including the baseline measurement. The exercise modalities include 1) continuous aerobic exercise, 2) high intensity exercise and 3) resistance exercise training. A set consists of test-retest of the same experiment.

The objectives of this pilot study are

1. to assess the longevity of the increased whole-body insulin sensitivity in the days following different exercise modalities
2. To estimate the intra-individual differences of different exercise modalities on whole-body insulin sensitivity the days following the last exercise bout
3. To assess the fidelity of the test- and exercise protocols

ELIGIBILITY:
Inclusion Criteria:

* BMI>25
* Age> 40 years
* Inactivity, defined as < 1,5 hours of structured physical activity pr. week at moderate intensity and cycling < 30 minutes/5 km pr. day at moderate intensity (moderate intensity = out of breath but able to speak)

Exclusion Criteria:

* • HbA1c>53 mmol/mol

  * Uncontrolled hypertension
  * Uncontrolled hyperlipidemia,
  * Known hyperthyroid disease
  * Endocrine disorders causing obesity
  * Known autoimmune disease
  * Unstable cardiovascular disease
  * Glucose lowering medications except for low dose metformin (=<1000 mg/day)
  * Current treatment with anti-inflammatory medication, unless pain killers without prescription
  * No participation in other research intervention studies
  * Pregnancy/considering pregnancy within the study period
  * Conditions countering exercise

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
24 hour change in insulin sensitivity (Matsuda index) derived from a 2-hour Oral Glucose Tolerance Test | 6 weeks
  Difference between exercise modalities in the change in whole-body insulin sensitivity (Matsuda index) from baseline to 24 hours following the exercise bout

SECONDARY OUTCOMES:
48 hour change in insulin sensitivity (Oral glucose insulin sensitivity index) derived from a 2-hour Oral Glucose Tolerance Test | 6 weeks
  Difference between exercise modalities in the change in whole-body insulin sensitivity (Oral glucose sensitivity index) from baseline to 48 hours following the exercise bout
24 hour change in insulin sensitivity (Oral glucose insulin sensitivity index) derived from a 2-hour Oral Glucose Tolerance Test | 6 weeks
  Difference between exercise modalities in the change in whole-body insulin sensitivity (Oral glucose insulin sensitivity index) from baseline to 24 hours following the exercise bout
48 hour change in insulin sensitivity (Matsuda index) derived from a 2-hour Oral Glucose Tolerance Test | 6 weeks
  Difference between exercise modalities in the change in whole-body insulin sensitivity (Matsuda index) from baseline to 48 hours following the exercise bout
24 to 48 hour change in insulin sensitivity (Oral glucose insulin sensitivity index) derived from a 2-hour Oral Glucose Tolerance Test | 6 weeks
  Difference between exercise modalities in the change in whole-body insulin sensitivity (Oral glucose sensitivity index) from 24 hours to 48 hours following the exercise bout
24 to 48 hour change in insulin sensitivity (Matsuda index) derived from a 2-hour Oral Glucose Tolerance Test | 6 weeks
  Difference between exercise modalities in the change in whole-body insulin sensitivity (Matsuda index) from 24 hours to 48 hours following the exercise bout
Variation in insulin sensitivity (Oral glucose sensitivity index) derived from a 2-hour Oral Glucose Tolerance Test | 6 weeks
  The typical difference between a pair of replicate measurements in whole-body insulin sensitivity (Oral glucose sensitivity index) in response to different exercise modalities 1 day following the previous exercise bout (intra-individual variation) and inter-individual response variability in whole-body insulin sensitivity (Oral glucose sensitivity index) in response to different exercise modalities 1 day following the previous exercise bout (inter-individual variation).
Variation in insulin sensitivity (Matsuda index) derived from a 2-hour Oral Glucose Tolerance Test | 6 weeks
  The typical difference between a pair of replicate measurements in whole-body insulin sensitivity (Matsuda index) in response to different exercise modalities 1 day following the previous exercise bout (intra-individual variation) and inter-individual response variability in whole-body insulin sensitivity (Matsuda index) in response to different exercise modalities 1 day following the previous exercise bout (inter-individual variation).
Variation in fasting and postprandial glucose | 6 weeks
  The typical difference between a pair of replicate measurements in fasting and post-prandial (derived from an OGTT) plasma glucose in response to different exercise modalities 1 day following the previous exercise bout (intra-individual variation) and inter-individual response variability in fasting and post-prandial (derived from an OGTT) plasma glucose in response to different exercise modalities 1 day following the previous exercise bout (inter-individual variation).
Variation in fasting and postprandial insulin | 6 weeks
  The typical difference between a pair of replicate measurements in fasting and post-prandial (derived from an OGTT) plasma insulin in response to different exercise modalities 1 day following the previous exercise bout (intra-individual variation) and inter-individual response variability in fasting and post-prandial (derived from an OGTT) plasma insulin in response to different exercise modalities 1 day following the previous exercise bout (inter-individual variation).
Variation in fasting and postprandial plasma C-peptide | 6 weeks
  The typical difference between a pair of replicate measurements in fasting and post-prandial (derived from an OGTT) plasma C-peptide in response to different exercise modalities 1 day following the previous exercise bout (intra-individual variation) and inter-individual response variability in fasting and post-prandial (derived from an OGTT) plasma C-peptide in response to different exercise modalities 1 day following the previous exercise bout (inter-individual variation).
Variation in gastric emptying | 6 weeks
  The typical difference between a pair of replicate measurements in post-prandial (from an OGTT) gastric empyting, measured by paracetamol, in response to different exercise modalities 1 day following the previous exercise bout (intra-individual variation) and inter-individual response variability in post-prandial (from an OGTT) gastric empyting, measured by paracetamol, in response to different exercise modalities 1 day following the previous exercise bout (inter-individual variation).
Assessment of free living physical activity | 6 weeks
  The typical difference between a pair of replicate measurements in free living physical activity (measured by accelerometers) in response to different exercise modalities 1 day following the previous exercise bout (intra-individual variation) and inter-individual response variability in free living physical activity (measured by accelerometers) in response to different exercise modalities 1 day following the previous exercise bout (inter-individual variation).
Assessment of continuous glucose | 6 weeks
  The typical difference between a pair of replicate measurements in continuous glucose (measured by continuous glucose monitors) in response to different exercise modalities following the previous exercise bout (intra-individual variation) and inter-individual response variability in continuous glucose (measured by continuous glucose monitors) in response to different exercise modalities following the previous exercise bout (inter-individual variation).
Assessment of psychosocial stress | 6 weeks
  The typical difference between a pair of replicate measurements in psychosocial stress (measured by questionnaires) in response to different exercise modalities following the previous exercise bout (intra-individual variation) and inter-individual response variability in psychosocial stress (measured by questionnaires) in response to different exercise modalities following the previous exercise bout (inter-individual variation).
Feasibility of the test and training protocols | 6 weeks
  Feasibility will be assessed using a qualitative questionnaires. Subject domains include e.g. participant satisfaction with 1) time spend on test- and training, 2) the recruitment process, 3) communication regarding participation and 4) the written information about participation, 5) acceptability of the tests.

CONTACTS AND LOCATIONS:
Overall Officials: Mathias Ried-Larsen, Ph D, Principal Investigator — Center for Physical Activity Research, Rigshospitalet
Locations (1):
- Center for Aktiv Sundhed - Rigshospitalet, Denmark (CFAS), Copenhagen, Østerbro, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
If the data can be fully anonymized the data can be shared.